CLINICAL TRIAL: NCT02994927
Title: A Randomized, Double-Blind, Active-Controlled, Phase 3 Study to Evaluate the Safety and Efficacy of CCX168 (Avacopan) in Patients With ANCA-Associated Vasculitis Treated Concomitantly With Rituximab or Cyclophosphamide/Azathioprine
Brief Title: A Phase 3 Clinical Trial of CCX168 (Avacopan) in Patients With ANCA-Associated Vasculitis
Acronym: ADVOCATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL010_168; ADVOCATE (Other: ChemoCentryx)
Record Dates: First submitted 2016-12-11; First posted 2016-12-16 (Estimated); Results first posted 2022-09-09 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: ANCA-Associated Vasculitis
Keywords: ANCA-associated vasculitis; complement; vasculitis; C5aR; avacopan; CCX168; MPA; GPA
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; Vasculitis | interventions — avacopan; Prednisone; Cyclophosphamide; Rituximab; Azathioprine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was double-blind, double-dummy, i.e., placebo capsules were identical in appearance to the avacopan capsules, and prednisone capsules also had matching placebo capsules. To maintain the blind, multiple measures were taken (i.e., randomization code was not accessible to study personnel who had contact with study centers or who were involved in data management and analysis for the duration of the study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prednisone group (Active Comparator): Avacopan-matching placebo plus cyclophosphamide/azathioprine or rituximab plus a full starting dose of prednisone.
  Interventions: Drug: Prednisone; Drug: Cyclophosphamide; Biological: Rituximab; Drug: Azathioprine
- Avacopan group (Experimental): Avacopan plus cyclophosphamide/azathioprine or rituximab plus prednisone-matching placebo.
  Interventions: Drug: Avacopan; Drug: Cyclophosphamide; Biological: Rituximab; Drug: Azathioprine

INTERVENTIONS:
Drug: Avacopan — Avacopan 30 mg twice daily orally for 52 weeks (364 days):
  - Three 10 mg avacopan capsules in the morning, preferably with food, and three in the evening, preferably with food, approximately 12 hours after the morning dose.
  Oral prednisone-matching placebo tapering regimen over 20 weeks (140 days):
  * Prednisone-matching placebo capsules equivalent to 60 mg per day if the subject's body weight was ≥55 kg, or 45 mg per day if the subject's body weight was <55 kg, starting on Day 1 with tapering according to a protocol-specified schedule.
  * Adolescents who weighed ≤37 kg started at a prednisone-matching placebo dose of 30 mg per day.
  Other Names: CCX168
  Arms: Avacopan group
Drug: Prednisone — Avacopan-matching placebo twice daily orally for 52 weeks (364 days):
  - Three avacopan-matching placebo capsules in the morning, preferably with food, and three in the evening, preferably with food, approximately 12 hours after the morning dose.
  Oral prednisone tapering regimen over 20 weeks (140 days):
  * Prednisone 60 mg per day if the subject's body weight was ≥55 kg, or 45 mg per day if the subject's body weight was <55 kg, starting on Day 1 with tapering according to the protocol-specified schedule.
  * Adolescents who weighed ≤37 kg started at a prednisone dose of 30 mg per day.
  Arms: Prednisone group
Drug: Cyclophosphamide — Orally or intravenously administered
Biological: Rituximab — Intravenously administered
Drug: Azathioprine — Orally administered

SUMMARY:
The primary objective is to evaluate the efficacy of CCX168 (avacopan) to induce and sustain remission in patients with active anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV), when used in combination with cyclophosphamide followed by azathioprine, or in combination with rituximab.

DETAILED DESCRIPTION:
Complement 5a and its receptor C5aR (CD88) are involved in the pathogenesis of anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis.

This is a randomized, double-blind, active-controlled Phase 3 study to evaluate the safety and efficacy of the orally-administered, selective C5aR inhibitor CCX168 (avacopan) in inducing and sustaining remission in patients with anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitis (AAV) treated concomitantly with Rituximab or Cyclophosphamide/Azathioprine.

Study acquired by Amgen and all disclosures were done by previous sponsor ChemoCentryx.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of granulomatosis with polyangiitis (Wegener's) or microscopic polyangiitis
* Male and female subjects, aged at least 18 years, with newly-diagnosed or relapsed associated vasculitis (AAV) where treatment with cyclophosphamide or rituximab is needed; where approved by Regulatory Agencies, adolescents (12-17 year old) may be enrolled
* Use of adequate contraception
* Positive test for anti-proteinase 3 (PR3) or anti-myeloperoxidase (MPO)
* At least 1 major item, or at least 3 non-major items, or at least the 2 renal items of proteinuria and hematuria on Birmingham Vasculitis Activity Score (BVAS)
* Estimated glomerular filtration rate ≥15 mL/minute/1.73 m^2 at screening

Exclusion Criteria:

* Pregnant or breast-feeding
* Alveolar hemorrhage requiring pulmonary ventilation support at screening
* Any other known multi-system autoimmune disease
* Required dialysis or plasma exchange within 12 weeks prior to screening
* Have a kidney transplant
* Received cyclophosphamide within 12 weeks prior to screening; if on azathioprine, mycophenolate mofetil or methotrexate at the time of screening, these drugs must be withdrawn prior to receiving the cyclophosphamide or rituximab dose on Day 1
* Received intravenous glucocorticoids, >3000 mg methylprednisolone equivalent, within 4 weeks prior to screening
* Have been taking an oral daily dose of a glucocorticoid of more than 10 mg prednisone-equivalent for more than 6 weeks continuously prior to screening
* Received rituximab or other B-cell antibody within 52 weeks of screening or 26 weeks provided B cell reconstitution has occurred (i.e., CD19 count > 0.01x10^9/L); received anti-tumor necrosis factor (TNF) treatment, abatacept, alemtuzumab, intravenous immunoglobulin (IVIg), belimumab, tocilizumab, or eculizumab within 12 weeks prior to screening
* For patients scheduled to receive cyclophosphamide treatment, urinary outflow obstruction, active infection (especially varicella zoster infection), or platelet count <50,000/μL before start of dosing
* Participated previously in a CCX168 study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2019-09-07 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (195):
- United States (38):
  - Clinical Trial Site, Huntsville, Alabama
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Santa Monica, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Daytona Beach, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Atlanta, Georgia
  - Clinical Trial Site, Meridian, Idaho
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Indianapolis, Indiana
  - Clinical Trial Site, Kansas City, Kansas
  - Clinical Trial Site, Lexington, Kentucky
  - Clinical Trial Site, Shreveport, Louisiana
  - Clinical Trial Site, Baltimore, Maryland
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Ann Arbor, Michigan
  - Clinical Trial Site, Minneapolis, Minnesota
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Great Neck, New York
  - Clinical Trial Site, Mineola, New York
  - Clinical Trial Site, New York, New York
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Greenville, North Carolina
  - Clinical Trial Site, Winston-Salem, North Carolina
  - Clinical Trial Site, Cleveland, Ohio
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Duncansville, Pennsylvania
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Providence, Rhode Island
  - Clinical Trial Site, Charleston, South Carolina
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
  - Clinical Trial Site, Salt Lake City, Utah
  - Clinical Trial Site, Seattle, Washington
- Australia (15):
  - Clinical Trial Site, Adelaide
  - Clinical Trial Site, Auchenflower
  - Clinical Trial Site, Brisbane
  - Clinical Trial Site, Clayton
  - Clinical Trial Site, Concord
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, Nambour
  - Clinical Trial Site, Nedlands
  - Clinical Trial Site, Randwick
  - Clinical Trial Site, Saint Albans
  - Clinical Trial Site, Southport
  - Clinical Trial Site, St Leonards
  - Clinical Trial Site, Westmead
  - Clinical Trial Site, Woolloongabba
- Austria (3):
  - Clinical Trial Site, Feldkirch
  - Clinical Trial Site, Graz
  - Clinical Trial Site, Innsbruck
- Belgium (4):
  - Clinical Trial Site, Antwerp
  - Clinical Trial Site, Brussels
  - Clinical Trial Site, Leuven
  - Clinical Trial Site, Liège
- Canada (8):
  - Clinical Trial Site, Calgary
  - Clinical Trial Site, Greenfield Park
  - Clinical Trial Site, Hamilton
  - Clinical Trial Site, Montreal
  - Clinical Trial Site, Québec
  - Clinical Trial Site, Sherbrooke
  - Clinical Trial Site, Toronto
  - Clinical Trial Site, Vancouver
- Czechia (2):
  - Clinical Trial Site, Olomouc
  - Clinical Trial Site, Prague
- Denmark (5):
  - Clinical Trial Site, Aalborg
  - Clinical Trial Site, Aarhus
  - Clinical Trial Site, Copenhagen
  - Clinical Trial Site, Odense
  - Clinical Trial Site, Roskilde
- France (15):
  - Clinical Trial Site, Angers
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Boulogne-sur-Mer
  - Clinical Trial Site, Brest
  - Clinical Trial Site, Bron
  - Clinical Trial Site, Caen
  - Clinical Trial Site, Colmar
  - Clinical Trial Site, Grenoble
  - Clinical Trial Site, Marseille
  - Clinical Trial Site, Metz
  - Clinical Trial Site, Nantes
  - Clinical Trial Site, Nîmes
  - Clinical Trial Site, Paris
  - Clinical Trial Site, Toulouse
  - Clinical Trial Site, Valenciennes
- Germany (20):
  - Clinical Trial Site, Aachen
  - Clinical Trial Site, Bad Bramstedt
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Cologne
  - Clinical Trial Site, Dresden
  - Clinical Trial Site, Essen
  - Clinical Trial Site, Freiburg im Breisgau
  - Clinical Trial Site, Fulda
  - Clinical Trial Site, Hamburg
  - Clinical Trial Site, Hanover
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Jena
  - Clinical Trial Site, Kirchheim unter Teck
  - Clinical Trial Site, Leipzig
  - Clinical Trial Site, Ludwigshafen
  - Clinical Trial Site, Lübeck
  - Clinical Trial Site, Mannheim
  - Clinical Trial Site, Munich
  - Clinical Trial Site, Tübingen
  - Clinical Trial Site, Villingen-Schwenningen
- Hungary (2):
  - Clinical Trial Site, Budapest
  - Clinical Trial Site, Debrecen
- Ireland (2):
  - Clinical Trial Site, Cork
  - Clinical Trial Site, Dublin
- Italy (9):
  - Clinical Trial Site, Ancona
  - Clinical Trial Site, Florence
  - Clinical Trial Site, Genova
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Monza
  - Clinical Trial Site, Parma
  - Clinical Trial Site, Reggio Emilia
  - Clinical Trial Site, Torino
  - Clinical Trial Site, Udine
- Japan (19):
  - Clinical Trial Site, Aichi
  - Clinical Trial Site, Akita
  - Clinical Trial Site, Chiba
  - Clinical Trial Site, Hiroshima
  - Clinical Trial Site, Hokkaido
  - Clinical Trial Site, Ishikawa
  - Clinical Trial Site, Kagawa
  - Clinical Trial Site, Kanagawa
  - Clinical Trial Site, Kobe
  - Clinical Trial Site, Miyazaki
  - Clinical Trial Site, Nagoya
  - Clinical Trial Site, Okayama
  - Clinical Trial Site, Osaka
  - Clinical Trial Site, Saitama
  - Clinical Trial Site, Shimane
  - Clinical Trial Site, Shizuoka
  - Clinical Trial Site, Tokyo
  - Clinical Trial Site, Toyama
  - Clinical Trial Site, Yokohama
- Netherlands (3):
  - Clinical Trial Site, Groningen
  - Clinical Trial Site, Leiden
  - Clinical Trial Site, Rotterdam
- New Zealand (5):
  - Clinical Trial Site, Christchurch
  - Clinical Trial Site, Dunedin
  - Clinical Trial Site, Grafton
  - Clinical Trial Site, Hamilton
  - Clinical Trial Site, Takapuna
- Norway (3):
  - Clinical Trial Site, Nordbyhagen
  - Clinical Trial Site, Oslo
  - Clinical Trial Site, Tromsø
- Spain (6):
  - Clinical Trial Site, Badalona
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Burela de Cabo
  - Clinical Trial Site, Lleida
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, San Sebastián
- Sweden (5):
  - Clinical Trial Site, Linköping
  - Clinical Trial Site, Lund
  - Clinical Trial Site, Örebro
  - Clinical Trial Site, Stockholm
  - Clinical Trial Site, Uppsala
- Switzerland (6):
  - Clinical Trial Site, Basel
  - Clinical Trial Site, Bern
  - Clinical Trial Site, Fribourg
  - Clinical Trial Site, Lausanne
  - Clinical Trial Site, Sankt Gallen
  - Clinical Trial Site, Zurich
- United Kingdom (25):
  - Clinical Trial Site, Aberdeen
  - Clinical Trial Site, Basildon
  - Clinical Trial Site, Birmingham
  - Clinical Trial Site, Bristol
  - Clinical Trial Site, Cambridge
  - Clinical Trial Site, Canterbury
  - Clinical Trial Site, Cardiff
  - Clinical Trial Site, Carshalton
  - Clinical Trial Site, Dorchester
  - Clinical Trial Site, Dudley
  - Clinical Trial Site, Exeter
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, Inverness
  - Clinical Trial Site, Kirkcaldy
  - Clinical Trial Site, Leeds
  - Clinical Trial Site, Leicester
  - Clinical Trial Site, Liverpool
  - Clinical Trial Site, London
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Newcastle
  - Clinical Trial Site, Nottingham
  - Clinical Trial Site, Oxford
  - Clinical Trial Site, Reading
  - Clinical Trial Site, Salford
  - Clinical Trial Site, Westcliff-on-Sea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- [Derived] Geetha D, Neumann T, Karras A, Cid MC, Merkel PA, Bray S, Bozeman AM, Jayne DRW; Members of the ADVOCATE Study Group. Efficacy and safety of avacopan for treatment of patients with ANCA-associated vasculitis receiving cyclophosphamide. RMD Open. 2025 Oct 5;11(4):e005743. doi: 10.1136/rmdopen-2025-005743. PMID 41052893
- [Derived] Geetha D, Dua A, Yue H, Springer J, Salvarani C, Jayne D, Merkel P; ADVOCATE Study Group. Efficacy and safety of avacopan in patients with ANCA-associated vasculitis receiving rituximab in a randomised trial. Ann Rheum Dis. 2024 Jan 11;83(2):223-232. doi: 10.1136/ard-2023-224816. PMID 37979959
- [Derived] Soulsby WD. Journal Club Review of "Avacopan for the Treatment of ANCA-Associated Vasculitis". ACR Open Rheumatol. 2022 Jul;4(7):558-561. doi: 10.1002/acr2.11412. Epub 2022 Feb 15. PMID 35167187
- [Derived] Jayne DRW, Merkel PA, Schall TJ, Bekker P; ADVOCATE Study Group. Avacopan for the Treatment of ANCA-Associated Vasculitis. N Engl J Med. 2021 Feb 18;384(7):599-609. doi: 10.1056/NEJMoa2023386. PMID 33596356
- [Derived] Merkel PA, Jayne DR, Wang C, Hillson J, Bekker P. Evaluation of the Safety and Efficacy of Avacopan, a C5a Receptor Inhibitor, in Patients With Antineutrophil Cytoplasmic Antibody-Associated Vasculitis Treated Concomitantly With Rituximab or Cyclophosphamide/Azathioprine: Protocol for a Randomized, Double-Blind, Active-Controlled, Phase 3 Trial. JMIR Res Protoc. 2020 Apr 7;9(4):e16664. doi: 10.2196/16664. PMID 32088663

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 143 study centers randomized at least 1 subject. The target enrollment was 300 subjects.
Pre-assignment Details: Screening details:
  Of 386 subjects screened, 331 were enrolled in the study and randomized to treatment. Reasons for subjects failing screening included not meeting inclusion/exclusion criteria, withdrawal by subject, adverse event (AE) and other.
Period: Overall Study
Arm/Group | Prednisone Group | Avacopan Group
Started | 165 | 166
Completed | 150 | 151
Not Completed | 15 | 15
Not completed — Withdrawal by parent/guardian | 0 | 1
Not completed — Did not meet eligibility criteria | 0 | 1
Not completed — Physician Decision | 4 | 3
Not completed — Death | 4 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 3 | 6
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Population: In the Prednisone group, one subject was randomized but withdrawn for not meeting disease criteria prior to dosing.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisone Group | Avacopan Group | Total
Number analyzed (Participants) | 164 | 166 | 330
Age, Customized [Count of Participants; unit: Participants]
  Adolescents (12-17 years) | 1 | 2 | 3
  Adults (18-50 years) | 28 | 30 | 58
  Adults (51-64 years) | 61 | 48 | 109
  Adults (65-75 years) | 52 | 62 | 114
  Adults (>75 years) | 22 | 24 | 46
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 68 | 144
  Male | 88 | 98 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 157 | 151 | 308
  Unknown or Not Reported | 2 | 8 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 17 | 32
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 140 | 138 | 278
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 6 | 8 | 14
Region of Enrollment [Number; unit: participants]
  Australia | 4 | 10 | 14
  Austria | 3 | 3 | 6
  Belgium | 4 | 6 | 10
  Canada | 5 | 8 | 13
  Czechia | 7 | 2 | 9
  Denmark | 10 | 6 | 16
  France | 18 | 22 | 40
  Germany | 32 | 22 | 54
  Italy | 2 | 9 | 11
  Japan | 10 | 11 | 21
  Netherlands | 5 | 1 | 6
  New Zealand | 2 | 2 | 4
  Ireland | 4 | 4 | 8
  Spain | 7 | 8 | 15
  Sweden | 2 | 5 | 7
  Switzerland | 6 | 4 | 10
  United Kingdom | 23 | 17 | 40
  United States | 20 | 26 | 46
Geographic Region [Count of Participants; unit: Participants]
  North America | 25 | 34 | 59
  Europe and Rest of World excluding Japan | 129 | 121 | 250
  Japan | 10 | 11 | 21
ANCA-associated vasculitis Status [Count of Participants; unit: Participants] — ANCA=anti-neutrophil cytoplasmic autoantibody
  Participants
    Newly diagnosed | 114 | 115 | 229
    Relapsed | 50 | 51 | 101
ANCA Positivity [Count of Participants; unit: Participants] — ANCA=anti-neutrophil cytoplasmic autoantibody
  Participants
    Proteinase 3 (PR3) | 70 | 72 | 142
    Myeloperoxidase (MPO) | 94 | 94 | 188
Standard of Care Treatment [Count of Participants; unit: Participants]
  Rituximab | 107 | 107 | 214
  Intravenous (IV) Cyclophosphamide | 51 | 51 | 102
  Oral Cyclophosphamide | 6 | 8 | 14
Type of ANCA-associated vasculitis [Count of Participants; unit: Participants] — ANCA=anti-neutrophil cytoplasmic autoantibody
  Participants
    Granulomatosis with polyangiitis (GPA) | 90 | 91 | 181
    Microscopic polyangiitis (MPA) | 74 | 75 | 149
BVAS Entry Criteria [Count of Participants; unit: Participants] — BVAS=Birmingham Vasculitis Activity Score;
  The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
  * Subjects can appear in more than one category
  Participants
    One or more major item | 102 | 104 | 206
    Three or more minor items | 142 | 146 | 288
    Two renal items of proteinuria and hematuria | 57 | 60 | 117
BVAS Components [Count of Participants; unit: Participants] — BVAS=Birmingham Vasculitis Activity Score
  * Subjects can appear in more than one category
  Participants
    General | 114 | 111 | 225
    Cutaneous | 23 | 24 | 47
    Mucous Membranes/Eyes | 40 | 26 | 66
    Ear Nose and Throat | 69 | 75 | 144
    Chest | 71 | 71 | 142
    Cardiovascular | 3 | 6 | 9
    Abdominal | 1 | 4 | 5
    Renal + Other (RBC Casts and/or Glomerulonephritis) | 134 | 134 | 268
    Nervous System | 31 | 38 | 69
Age at screening [Mean (Standard Deviation); unit: years] | 60.5 (14.50) | 61.2 (14.56) | 60.9 (14.51)
Age at diagnosis of ANCA-associated Vasculitis [Mean (Standard Deviation); unit: years] — ANCA=anti-neutrophil cytoplasmic autoantibody
  years | 59.4 (15.19) | 59.8 (15.60) | 59.6 (15.37)
Duration of ANCA-Associated Vasculitis [Mean (Standard Deviation); unit: months] — ANCA=anti-neutrophil cytoplasmic autoantibody
  months | 20.13 (40.473) | 22.93 (52.464) | 21.54 (46.840)
Body Weight [Mean (Standard Deviation); unit: kilogram(s)] | 77.71 (19.335) | 76.43 (20.254) | 77.07 (19.783)
BMI [Mean (Standard Deviation); unit: kilogram(s)/square meter] — BMI=Body Mass Index Population: Two subjects did not have a baseline BMI provided (one in each treatment group)
  kilogram(s)/square meter
    number analyzed (Participants) | 163 | 165 | 328
    (all) | 26.78 (5.212) | 26.72 (5.997) | 26.75 (5.612)
BVAS Score [Mean (Standard Deviation); unit: units on a scale] — BVAS=Birmingham Vasculitis Activity Score; The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
  units on a scale | 16.2 (5.69) | 16.3 (5.87) | 16.2 (5.77)
VDI Score [Mean (Standard Deviation); unit: units on a scale] — VDI=Vasculitis Damage Index; The VDI is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health). Population: Two subjects did not have a baseline VDI Score (one in each treatment group)
  units on a scale
    number analyzed (Participants) | 163 | 165 | 328
    (all) | 0.7 (1.39) | 0.7 (1.54) | 0.7 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Achieving Disease Remission at Week 26
Description: Disease remission at Week 26 was defined as:
  * Achieving a BVAS of 0 as determined by the Adjudication Committee;
  * No administration of glucocorticoids given for ANCA-associated vasculitis within 4 weeks prior to Week 26;
  * No BVAS >0 during the 4 weeks prior to Week 26 (if collected for an unscheduled assessment).
Time Frame: Week 26
Population: Intent-to-Treat (ITT) Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
percentage of participants | 70.1 [62.5 to 77.0] | 72.3 [64.8 to 78.9]
Statistical Analysis 1: Comparison: Prednisone Group vs Avacopan Group; Test type: Non-Inferiority — The proportion of subjects achieving disease remission at Week 26 and the two-sided 95% confidence intervals (CIs) for the difference in proportions was estimated for the comparison between the avacopan group and the prednisone group. For both the noninferiority and superiority tests, the one-sided P-values are presented. Statistical significance was claimed based on the one-sided type-I error of 0.025; p < 0.0001, Summary score test; Common difference in remission rates = 3.4, 95% CI 2-sided [-6.0 to 12.8] — Summary Score estimate of the common difference and Miettinen-Nurminen (score) confidence limits for the common difference
Statistical Analysis 2: Comparison: Prednisone Group vs Avacopan Group; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.2387, Summary score test; Common difference in remission rates = 3.4, 95% CI 2-sided [-6.0 to 12.8] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Percentage of Subjects Achieving Sustained Disease Remission at Week 52
Description: Sustained remission at Week 52 was defined as:
  * Disease remission at Week 26 as defined above;
  * Disease remission at Week 52 defined as a BVAS of 0 at Week 52 as determined by the Adjudication Committee and no administration of glucocorticoids for treatment of ANCA-associated vasculitis within 4 weeks prior to Week 52;
  * No disease relapse between Week 26 and Week 52 as determined by the Adjudication Committee.
Time Frame: Week 52
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
percentage of participants | 54.9 [46.9 to 62.6] | 65.7 [57.9 to 72.8]
Statistical Analysis 1: Comparison: Prednisone Group vs Avacopan Group; Test type: Non-Inferiority — The proportion of subjects achieving sustained disease remission at Week 52, and the two-sided 95% confidence intervals (CIs) for the difference in proportions (avacopan minus prednisone) was estimated for the comparison between the avacopan group and the prednisone group. For both the noninferiority and superiority tests, the one-sided P-values are presented. Statistical significance was claimed based on the one-sided type-I error of 0.025; p < 0.0001, Summary score test; Common difference in remission rates = 12.5, 95% CI 2-sided [2.6 to 22.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Prednisone Group vs Avacopan Group; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p = 0.0066, Summary score test; Common difference in remission rates = 12.5, 95% CI 2-sided [2.6 to 22.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Subject Incidence of Treatment-emergent SAEs, AEs, and Withdrawals Due to AEs
Description: AEs=Adverse events
  SAEs=Serious adverse events
  TEAE=Treatment-emergent adverse event
Time Frame: From day 1 throughout the study period (day 421/week 60)
Population: Safety Population: The safety population included all subjects who were randomized and had received at least one dose of study drug.
Measure: Number; unit: Number
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
Number
  Number of subjects with at least one TEAE | 161 | 164
  Number of TEAEs | 2139 | 1779
  Number of subjects with SAEs | 74 | 70
  Number of SAEs | 166 | 116
  Subjects with TEAE leading to discontinuation | 28 | 27

4. Secondary Outcome: Glucocorticoid-induced Toxicity as Measured by Change From Baseline Over the First 26 Weeks in the GTI
Description: GTI-CWS=Glucocorticoid Toxicity Index Cumulative Worsening Score;
  GTI-AIS=Glucocorticoid Toxicity Index Aggregate Improvement Score;
  The Glucocorticoid Toxicity Index (GTI) was developed to score glucocorticoid toxicity. The GTI includes: the Cumulative Worsening Score (CWS) that captures cumulative toxicity, both permanent and transient, over the course of time (serves as a cumulative record of toxicity); and the Aggregate Improvement Score that captures both improvement and worsening of toxicity over time (serves as a record of both improving and worsening toxicity). Both scores range from 0 (best health) to 100 (worst health).
Time Frame: Baseline, Week 13 and 26
Population: Intent-to-Treat (ITT) Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug. The number of subjects with data at the specified visit is reported.
Measure: Least Squares Mean (Standard Error); unit: Glucocorticoid Toxicity Index
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
Glucocorticoid Toxicity Index
  GTI-CWS (Week 13): number analyzed (Participants) | 161 | 160
  GTI-CWS (Week 13) | 36.6 (3.41) | 25.7 (3.40)
  GTI-CWS (Week 26): number analyzed (Participants) | 153 | 154
  GTI-CWS (Week 26) | 56.6 (3.45) | 39.7 (3.43)
  GTI-AIS (Week 13): number analyzed (Participants) | 161 | 160
  GTI-AIS (Week 13) | 23.2 (3.46) | 9.9 (3.45)
  GTI-AIS (Week 26): number analyzed (Participants) | 153 | 154
  GTI-AIS (Week 26) | 23.4 (3.50) | 11.2 (3.48)

5. Secondary Outcome: Percentage of Participants With BVAS of 0 at Week 4, Regardless of Whether the Subjects Received Glucocorticoids During This Period of Time and Based on Assessment by the Blinded AC
Description: AC=Adjudication Committee; BVAS=Birmingham Vasculitis Activity Score;
  The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
Time Frame: Week 4
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
percentage of participants | 68.9 [61.2 to 75.9] | 62.7 [54.8 to 70.0]

6. Secondary Outcome: Change From Baseline Over 52 Weeks in Health-related Quality of Life as Measured by the Domains and Component Scores of the SF-36v2 and EQ-5D-5L VAS and Index
Description: SF-36v2: Measure of health- related quality of life (Medical Outcomes Survey Short Form-36 version 2)
  EQ-5D-5L: EuroQuality of Life-5 Domains-5 Levels
  The SF-36v2 component scores and the EQ-5D-5L VAS score range from 0 (worst health) to 100 (best health). The EQ-5D-5L Index Score ranges from 0 (worst health) to 1 (best health).
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: Change from baseline
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 150 | 154
Change from baseline
  SF-36v2: Physical Component Score (Week 26): number analyzed (Participants) | 147 | 153
  SF-36v2: Physical Component Score (Week 26) | 1.344 (0.7432) | 4.445 (0.7332)
  SF-36v2: Physical Component Score (Week 52): number analyzed (Participants) | 144 | 147
  SF-36v2: Physical Component Score (Week 52) | 2.626 (0.7505) | 4.980 (0.7435)
  SF-36v2: Physical Functioning (Week 26): number analyzed (Participants) | 150 | 153
  SF-36v2: Physical Functioning (Week 26) | 1.88 (1.787) | 7.31 (1.773)
  SF-36v2: Physical Functioning (Week 52): number analyzed (Participants) | 145 | 149
  SF-36v2: Physical Functioning (Week 52) | 4.82 (1.809) | 9.55 (1.790)
  SF-36v2: Role Physical (Week 26) | 7.52 (2.198) | 16.78 (2.173)
  SF-36v2: Role Physical (Week 52): number analyzed (Participants) | 145 | 150
  SF-36v2: Role Physical (Week 52) | 12.27 (2.228) | 17.12 (2.198)
  SF-36v2: Bodily Pain (Week 26): number analyzed (Participants) | 149 | 154
  SF-36v2: Bodily Pain (Week 26) | 9.82 (2.197) | 14.75 (2.164)
  SF-36v2: Bodily Pain (Week 52): number analyzed (Participants) | 145 | 150
  SF-36v2: Bodily Pain (Week 52) | 11.87 (2.220) | 16.12 (2.185)
  SF-36v2: General Health Perception (Week 26): number analyzed (Participants) | 148 | 154
  SF-36v2: General Health Perception (Week 26) | -2.89 (1.428) | 3.12 (1.405)
  SF-36v2: General Health Perception (Week 52): number analyzed (Participants) | 145 | 150
  SF-36v2: General Health Perception (Week 52) | -0.17 (1.442) | 5.84 (1.420)
  SF-36v2: Mental Component Score (Week 26): number analyzed (Participants) | 147 | 154
  SF-36v2: Mental Component Score (Week 26) | 3.271 (0.8403) | 4.849 (0.8273)
  SF-36v2: Mental Component Score (Week 52): number analyzed (Participants) | 144 | 148
  SF-36v2: Mental Component Score (Week 52) | 4.694 (0.8491) | 6.394 (0.8406)
  SF-36v2: Mental Health (Week 26): number analyzed (Participants) | 148 | 154
  SF-36v2: Mental Health (Week 26) | 6.84 (1.331) | 8.29 (1.318)
  SF-36v2: Mental Health (Week 52): number analyzed (Participants) | 144 | 148
  SF-36v2: Mental Health (Week 52) | 9.66 (1.347) | 10.89 (1.337)
  SF-36v2: Role Emotional (Week 26) | 1.40 (2.183) | 7.32 (2.158)
  SF-36v2: Role Emotional (Week 52): number analyzed (Participants) | 145 | 150
  SF-36v2: Role Emotional (Week 52) | 4.14 (2.212) | 9.38 (2.181)
  SF-36v2: Social Functioning (Week 26): number analyzed (Participants) | 147 | 154
  SF-36v2: Social Functioning (Week 26) | 11.09 (2.037) | 14.50 (2.002)
  SF-36v2: Social Functioning (Week 52): number analyzed (Participants) | 144 | 149
  SF-36v2: Social Functioning (Week 52) | 13.56 (2.059) | 18.06 (2.030)
  SF-36v2: Vitality (Week 26): number analyzed (Participants) | 148 | 154
  SF-36v2: Vitality (Week 26) | 6.42 (1.751) | 12.03 (1.727)
  SF-36v2: Vitality (Week 52): number analyzed (Participants) | 144 | 148
  SF-36v2: Vitality (Week 52) | 10.48 (1.770) | 14.36 (1.750)
  EQ-5D-5L VAS Score (Week 26): number analyzed (Participants) | 150 | 153
  EQ-5D-5L VAS Score (Week 26) | 5.5 (1.39) | 9.1 (1.38)
  EQ-5D-5L VAS Score (Week 52): number analyzed (Participants) | 146 | 149
  EQ-5D-5L VAS Score (Week 52) | 7.1 (1.41) | 13.0 (1.39)
  EQ-5D-5L Index Score (Week 26): number analyzed (Participants) | 146 | 152
  EQ-5D-5L Index Score (Week 26) | -0.0010 (0.01462) | 0.0229 (0.01438)
  EQ-5D-5L Index Score (Week 52): number analyzed (Participants) | 145 | 149
  EQ-5D-5L Index Score (Week 52) | -0.0038 (0.01471) | 0.0474 (0.01451)

7. Secondary Outcome: Percentage of Subjects and Time to Experiencing a Relapse After Previously Achieving Remission at Week 26 in the Study
Description: The median time to relapse was not estimable because of small number of relapsed subjects.
  A relapse was defined as occurrence of at least one major item in the BVAS, or three or more minor items in the BVAS, or one or two minor items in the BVAS recorded at two consecutive visits, after:
  1. having achieved remission at Week 26 (BVAS=0 and no glucocorticoids for ANCA-associated vasculitis within 4 weeks) or
  2. having achieved BVAS=0 at any time during the treatment period
  ANCA=anti-neutrophil cytoplasmic autoantibody; BVAS=Birmingham Vasculitis Activity Score; The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
Time Frame: Week 52
Population: Intent-to-Treat (ITT) Subjects in the analysis population for the specified treatment group.
  ITT Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 115 | 120
percentage of participants | 12.2 [6.8 to 19.6] | 7.5 [3.5 to 13.8]

8. Secondary Outcome: Percentage of Subjects and Time to Experiencing a Relapse After Previously Achieving BVAS=0 at Any Time During the Treatment Period
Description: The median time to relapse was not estimable because of small number of relapsed subjects.
  A relapse was defined as occurrence of at least one major item in the BVAS, or three or more minor items in the BVAS, or one or two minor items in the BVAS recorded at two consecutive visits, after:
  1. having achieved remission at Week 26 (BVAS=0 and no glucocorticoids for ANCA-associated vasculitis within 4 weeks) or
  2. having achieved BVAS=0 at any time during the treatment period
  The Birmingham Vasculitis Activity Score (BVAS) form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
Time Frame: Week 52
Population: Intent-to-Treat (ITT) Subjects who achieved BVAS=0 during the 52 week treatment period.
  ITT Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 157 | 158
percentage of participants | 21.0 [14.9 to 28.2] | 10.1 [5.9 to 15.9]

9. Secondary Outcome: In Subjects With Renal Disease at Baseline (Based in the BVAS Renal Component), the Change in eGFR From Baseline Over 52 Weeks
Description: Change from baseline in kidney function, as measured by eGFR (based on the MDRD equation), was measured in subjects with renal disease based on the BVAS renal component.
  eGFR=estimated glomerular filtration rate
  BVAS=Birmingham Vasculitis Activity Score
  MDRD=Modification of Diet in Renal Disease
Time Frame: Baseline, Week 26 and 52
Population: Intent-to-Treat (ITT) Subjects With Renal Disease at Baseline (based on BVAS).
  ITT Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in eGFR (mL/min/1.73 m^2)
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 127 | 121
Change in eGFR (mL/min/1.73 m^2)
  Week 26 | 2.9 [0.9 to 4.9] | 5.8 [3.7 to 7.8]
  Week 52: number analyzed (Participants) | 125 | 119
  Week 52 | 4.1 [2.1 to 6.1] | 7.3 [5.2 to 9.4]

10. Secondary Outcome: In Subjects With Renal Disease and Albuminuria at Baseline (Based in the BVAS Renal Component), the Percent Change in UACR From Baseline Over 52 Weeks
Description: BVAS=Birmingham Vasculitis Activity Score
  UACR=Urinary albumin:creatinine ratio
Time Frame: Baseline, Week 4, 26 and 52
Population: Intent-to-Treat (ITT) Subjects With Renal Disease (based on BVAS) and Albuminuria (UACR>=10 mg/g creatinine) at Baseline
  ITT Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 124 | 121
Percentage change
  Week 4 | 0 [-16 to 19] | -40 [-50 to -28]
  Week 26: number analyzed (Participants) | 118 | 113
  Week 26 | -70 [-75 to -65] | -63 [-69 to -56]
  Week 52: number analyzed (Participants) | 114 | 109
  Week 52 | -77 [-81 to -72] | -74 [-78 to -69]

11. Secondary Outcome: In Subjects With Renal Disease at Baseline (Based in the BVAS Renal Component), the Percent Change in Urinary MCP-1:Creatinine Ratio From Baseline Over 52 Weeks
Description: BVAS=Birmingham Vasculitis Activity Score
  MCP-1=monocyte chemoattractant protein-1
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage change
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 117 | 106
Percentage change
  Week 26 | -64 [-67 to -59] | -67 [-70 to -63]
  Week 52: number analyzed (Participants) | 108 | 106
  Week 52 | -71 [-74 to -67] | -73 [-76 to -70]

12. Secondary Outcome: Change in the VDI From Baseline Over 52 Weeks, Including the Week 26 and Week 52 Time Points
Description: VDI=Vasculitis Damage Index; The VDI is comprised of 64 items of damage, grouped into 11 organ-based systems or categorizations. Damage is defined as the presence of non-healing scars and does not give any indication of current disease activity. Damage is also defined as having been present or currently present for at least 3 months. Completion of the form provides a numerical score, which ranges from 0 (best health) to 64 (worst health).
Time Frame: Baseline, Week 26 and 52
Population: Intent-to-Treat (ITT) Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug. The number of subjects with data at baseline and the specified visit is reported.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 155 | 161
score on a scale
  Week 26 | 0.97 (0.092) | 1.06 (0.090)
  Week 52: number analyzed (Participants) | 151 | 150
  Week 52 | 1.15 (0.093) | 1.17 (0.091)

13. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Hematology (1/5)
Time Frame: Baseline, Week 26 and 52
Population: Safety Population: The safety population included all subjects who were randomized and had received at least one dose of study drug. The number of subjects with data at baseline and the specified visit is reported.
Measure: Mean (Standard Error); unit: 10^3 cells/μL
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 151 | 147
10^3 cells/μL
  Leukocytes (Week 26) | -5.69 (0.338) | -5.94 (0.387)
  Leukocytes (Week 52): number analyzed (Participants) | 149 | 147
  Leukocytes (Week 52) | -5.54 (0.365) | -5.62 (0.395)
  Neutrophils (Week 26): number analyzed (Participants) | 148 | 143
  Neutrophils (Week 26) | -5.10 (0.338) | -5.24 (0.380)
  Neutrophils (Week 52): number analyzed (Participants) | 147 | 144
  Neutrophils (Week 52) | -4.89 (0.361) | -4.95 (0.372)
  Lymphocytes (Week 26): number analyzed (Participants) | 148 | 143
  Lymphocytes (Week 26) | -0.62 (0.090) | -0.84 (0.099)
  Lymphocytes (Week 52): number analyzed (Participants) | 147 | 144
  Lymphocytes (Week 52) | -0.67 (0.090) | -0.82 (0.100)

14. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Hematology (2/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: 10^9 cells/L
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 147
10^9 cells/L
  Eosinophils (Week 26): number analyzed (Participants) | 148 | 143
  Eosinophils (Week 26) | 0.07 (0.016) | 0.07 (0.018)
  Eosinophils (Week 52): number analyzed (Participants) | 147 | 144
  Eosinophils (Week 52) | 0.05 (0.013) | 0.07 (0.019)
  Basophils (Week 26): number analyzed (Participants) | 148 | 143
  Basophils (Week 26) | -0.01 (0.004) | -0.00 (0.004)
  Basophils (Week 52): number analyzed (Participants) | 147 | 144
  Basophils (Week 52) | -0.01 (0.004) | -0.01 (0.004)
  Monocytes (Week 26): number analyzed (Participants) | 148 | 143
  Monocytes (Week 26) | 0.01 (0.022) | -0.04 (0.024)
  Monocytes (Week 52): number analyzed (Participants) | 147 | 144
  Monocytes (Week 52) | 0.01 (0.024) | -0.01 (0.026)
  Platelets (Week 26) | -73.9 (8.49) | -77.1 (9.30)
  Platelets (Week 52): number analyzed (Participants) | 149 | 146
  Platelets (Week 52) | -75.5 (8.01) | -73.8 (9.31)

15. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Hematology (3/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: 10^12 cells/L
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 147
10^12 cells/L
  Erythrocytes (Week 26) | 0.226 (0.0450) | 0.252 (0.0432)
  Erythrocytes (Week 52): number analyzed (Participants) | 149 | 147
  Erythrocytes (Week 52) | 0.244 (0.0410) | 0.279 (0.0432)

16. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Hematology (4/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 147
g/dL
  Hemoglobin (Week 26) | 1.07 (0.129) | 1.10 (0.120)
  Hemoglobin (Week 52): number analyzed (Participants) | 149 | 147
  Hemoglobin (Week 52) | 1.20 (0.126) | 1.27 (0.125)

17. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Hematology (5/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: percentage of red blood cells
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 147
percentage of red blood cells
  Hematocrit (Week 26) | 2.6 (0.38) | 2.7 (0.38)
  Hematocrit (Week 52): number analyzed (Participants) | 149 | 147
  Hematocrit (Week 52) | 3.0 (0.37) | 3.2 (0.38)

18. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Serum Chemistry (1/2)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 154 | 150
U/L
  Lactate Dehydrogenase (Week 26): number analyzed (Participants) | 149 | 145
  Lactate Dehydrogenase (Week 26) | 2.3 (5.68) | -6.1 (5.40)
  Lactate Dehydrogenase (Week 52): number analyzed (Participants) | 146 | 141
  Lactate Dehydrogenase (Week 52) | -8.6 (5.33) | -10.7 (4.80)
  Alkaline Phosphatase (Week 26) | -0.6 (2.47) | -3.9 (2.84)
  Alkaline Phosphatase (Week 52): number analyzed (Participants) | 152 | 147
  Alkaline Phosphatase (Week 52) | 0.8 (1.77) | -4.0 (2.34)
  Creatine Kinase (Week 26) | 47.6 (5.27) | 76.8 (10.34)
  Creatine Kinase (Week 52): number analyzed (Participants) | 152 | 147
  Creatine Kinase (Week 52) | 57.6 (5.67) | 76.3 (9.68)
  Alanine Aminotransferase (Week 26) | -6.8 (1.77) | -6.1 (1.54)
  Alanine Aminotransferase (Week 52): number analyzed (Participants) | 152 | 147
  Alanine Aminotransferase (Week 52) | -8.2 (1.57) | -7.2 (1.46)
  Aspartate Aminotransferase (Week 26) | 1.9 (0.98) | 2.5 (0.72)
  Aspartate Aminotransferase (Week 52): number analyzed (Participants) | 152 | 147
  Aspartate Aminotransferase (Week 52) | 0.5 (0.85) | 2.0 (0.69)

19. Secondary Outcome: Change From Baseline and Shifts From Baseline in All Safety Laboratory Parameters - Serum Chemistry (2/2)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 159 | 162
mg/dL
  Creatinine (Week 26): number analyzed (Participants) | 154 | 150
  Creatinine (Week 26) | -0.105 (0.0569) | -0.195 (0.0508)
  Creatinine (Week 52): number analyzed (Participants) | 152 | 147
  Creatinine (Week 52) | -0.200 (0.0416) | -0.244 (0.0627)
  Urea Nitrogen (Week 26): number analyzed (Participants) | 154 | 150
  Urea Nitrogen (Week 26) | -9.4 (1.16) | -11.0 (1.32)
  Urea Nitrogen (Week 52): number analyzed (Participants) | 152 | 147
  Urea Nitrogen (Week 52) | -7.8 (1.11) | -11.9 (1.32)
  Protein (Week 26): number analyzed (Participants) | 154 | 150
  Protein (Week 26) | 50 (50) | 220 (47)
  Protein (Week 52): number analyzed (Participants) | 152 | 147
  Protein (Week 52) | 160 (48) | 250 (41)
  Cholesterol (Week 26): number analyzed (Participants) | 154 | 150
  Cholesterol (Week 26) | 19.0 (4.27) | 7.4 (3.99)
  Cholesterol (Week 52): number analyzed (Participants) | 152 | 147
  Cholesterol (Week 52) | 13.8 (4.28) | 9.3 (4.05)
  LDL Cholesterol (Week 26): number analyzed (Participants) | 154 | 152
  LDL Cholesterol (Week 26) | 22.7 (3.66) | 12.0 (3.47)
  LDL Cholesterol (Week 52) | 21.7 (3.48) | 11.9 (3.41)
  Bilirubin (Week 26): number analyzed (Participants) | 154 | 150
  Bilirubin (Week 26) | 0.065 (0.0182) | 0.078 (0.0250)
  Bilirubin (Week 52): number analyzed (Participants) | 152 | 147
  Bilirubin (Week 52) | 0.053 (0.0185) | 0.057 (0.0201)

20. Secondary Outcome: Change From Baseline in Vital Signs (1/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 154 | 154
mmHg
  Systolic Blood Pressure (Week 26) | -2.5 (1.70) | -2.6 (1.54)
  Systolic Blood Pressure (Week 52): number analyzed (Participants) | 151 | 150
  Systolic Blood Pressure (Week 52) | -2.4 (1.64) | -1.0 (1.60)
  Diastolic Blood Pressure (Week 26) | 2.7 (0.98) | 0.5 (0.92)
  Diastolic Blood Pressure (Week 52): number analyzed (Participants) | 151 | 150
  Diastolic Blood Pressure (Week 52) | 1.4 (1.01) | 1.4 (1.00)

21. Secondary Outcome: Change From Baseline in Vital Signs (2/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: beats/min
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 154
beats/min
  Pulse Rate (Week 26) | 2.2 (1.12) | 0.9 (1.25)
  Pulse Rate (Week 52): number analyzed (Participants) | 151 | 150
  Pulse Rate (Week 52) | -1.3 (1.07) | -0.3 (1.21)

22. Secondary Outcome: Change From Baseline in Vital Signs (3/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: degree Celsius
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 152 | 151
degree Celsius
  Temperature (Week 26) | -0.03 (0.043) | -0.11 (0.046)
  Temperature (Week 52): number analyzed (Participants) | 148 | 148
  Temperature (Week 52) | 0.04 (0.044) | -0.11 (0.048)

23. Secondary Outcome: Change From Baseline in Vital Signs (4/5)
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: kilogram(s)
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 154 | 153
kilogram(s)
  Weight (Week 26) | 3.33 (0.397) | 1.93 (0.369)
  Weight (Week 52): number analyzed (Participants) | 151 | 150
  Weight (Week 52) | 3.27 (0.477) | 2.59 (0.487)

24. Secondary Outcome: Change From Baseline in Vital Signs (5/5)
Description: BMI=Body Mass Index
Time Frame: Baseline, Week 26 and 52
Population: as for outcome 13
Measure: Mean (Standard Error); unit: kilogram(s)/ square meter
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 153 | 152
kilogram(s)/ square meter
  BMI (Week 26) | 1.13 (0.135) | 0.67 (0.132)
  BMI (Week 52): number analyzed (Participants) | 150 | 149
  BMI (Week 52) | 1.12 (0.164) | 0.94 (0.179)

25. Secondary Outcome: Number of Subjects With Clinically Significant ECG Changes From Baseline
Description: Clinical significance was assessed by the individual reading of the ECGs
  ECG=Electrocardiogram
Time Frame: From day 1 throughout the study period (day 421/week 60)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
Participants | 8 | 12

26. Secondary Outcome: Number of Subjects Where a Relationship Between Avacopan/Placebo, Glucocorticoid Use, Cyclophosphamide, Rituximab, and Azathioprine or Mycophenolate Use to an AE Was Determined by the Investigator
Description: AE=Adverse Event
Time Frame: From day 1 throughout the study period (day 421/week 60)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
Participants
  Relationship of avacopan/placebo to an AE | 103 | 100
  Relationship of glucocorticoid use to an AE | 131 | 107
  Relationship of cyclophosphamide IV use to an AE | 30 | 31
  Relationship of oral cyclophosphamide use to an AE | 4 | 8
  Relationship of rituximab use to an AE | 61 | 50
  Relationship of azathioprine use to an AE | 35 | 28
  Relationship of mycophenolate use to an AE | 9 | 6

27. Secondary Outcome: Certain Safety Endpoints of Interest: Infections, Hepatic System Abnormalities, WBC Count Decreases, and Hypersensitivity
Description: WBC=White Blood Cell
  TEAE=Treatment-Emergent Adverse Event
Time Frame: From day 1 throughout the study period (day 421/week 60)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 164 | 166
Participants
  Any Treatment-Emergent Infection | 124 | 113
  Any Serious Treatment-Emergent Infection | 25 | 22
  Any Severe Treatment-Emergent Infection | 10 | 12
  Any Treatment-Emergent Infection Leading to Study Withdrawal | 5 | 4
  Any Treatment-Emergent Life-threatening Infection | 2 | 1
  Any Treatment-Emergent Infection Leading to Death | 2 | 1
  Any TEAE Associated with Hepatic Abnormalities | 19 | 22
  Any TEAE Associated with Low WBC Counts | 39 | 31
  Any TEAE Associated with hypersensitivity | 70 | 68

28. Secondary Outcome: Number of Subjects Experiencing a Relapse After Previously Achieving BVAS=0 During the Study
Description: BVAS=Birmingham Vasculitis Activity Score;
  A relapse was defined as occurrence of at least one major item in the BVAS, or three or more minor items in the BVAS, or one or two minor items in the BVAS recorded at two consecutive visits, after:
  1. having achieved remission at Week 26 (BVAS=0 and no glucocorticoids for ANCA-associated vasculitis within 4 weeks) or
  2. having achieved BVAS=0 at any time during the treatment period
  The BVAS form is divided into 9 organ-based systems, with each section including symptoms/signs that are typical of that particular organ involvement in systemic vasculitis. The clinician only scores features believed to be due to active vasculitis. Completion of the form provides a numerical score, which ranges from 0 (best health) to 63 (worst health).
Time Frame: From day 1 throughout the study period (day 421/week 60)
Population: Intended-to-Treat (ITT) Population: The ITT Population included all subjects who were randomized in the study and who received at least one dose of blinded study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone Group | Avacopan Group
Number analyzed (Participants) | 157 | 158
Participants | 33 | 16

ADVERSE EVENTS:
Time Frame: From day 1 throughout the study period (day 421/week 60)
Description: An AE was considered treatment-emergent if the start date/time of the event was on or after the date/time of first dose of study drug through 56 days following the last dose administered during the randomized treatment period.
Groups:
- Prednisone Group: Avacopan-matching placebo plus cyclophosphamide/azathioprine or rituximab plus a full starting dose of prednisone. The safety population included all subjects who were randomized and had received at least one dose of study drug.
- Avacopan Group: Avacopan plus cyclophosphamide/azathioprine or rituximab plus prednisone-matching placebo. The safety population included all subjects who were randomized and had received at least one dose of study drug.
Arm/Group | Prednisone Group | Avacopan Group
All-Cause Mortality (participants affected / at risk) | 4/164 | 2/166
Serious Adverse Events (participants affected / at risk) | 74/164 | 70/166
Other Adverse Events (participants affected / at risk) | 161/164 | 164/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone Group (N=164) | Avacopan Group (N=166)
Granulomatosis with polyangiitis (Vascular disorders) | 1 (1) | 5 (5)
Microscopic polyangiitis (Vascular disorders) | 2 (2) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 2 (3) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 2 (3)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 20 (25) | 12 (12)
Hepatic enzyme increased (Investigations) | 3 (3) | 2 (2)
Blood creatinine increased (Investigations) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Agranulocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Mononeuropathy multiplex (Nervous system disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 3 (3)
Glomerulonephritis (Renal and urinary disorders) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 6 (6) | 8 (9)
Urinary tract infection (Infections and infestations) | 2 (2) | 3 (3)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2)
Herpes zoster (Infections and infestations) | 2 (2) | 0 (0)
Infectious pleural effusion (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 2 (2) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 2 (2) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Antineutrophil cytoplasmic antibody increased (Investigations) | 0 (0) | 1 (1)
Arteriovenous fistula operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia haemophilus (Infections and infestations) | 0 (0) | 1 (1)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Aspergillus infection (Infections and infestations) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone marrow toxicity (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Cryptococcosis (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Episcleritis (Eye disorders) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Granulomatous lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Medical observation (Investigations) | 1 (1) | 0 (0)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nervous system disorder (Nervous system disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Ophthalmic herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngeal ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone Group (N=164) | Avacopan Group (N=166)
Hypertension (Vascular disorders) | 29 (31) | 30 (36)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 34 (46) | 26 (30) — Worsening of vasculitis is reported as the Preferred Term of "anti-neutrophil cytoplasmic antibody-positive vasculitis".
Oedema peripheral (General disorders) | 40 (56) | 35 (39)
Fatigue (General disorders) | 15 (15) | 17 (19)
Pyrexia (General disorders) | 19 (25) | 15 (18)
Insomnia (Psychiatric disorders) | 25 (27) | 13 (13)
Weight increased (Investigations) | 17 (19) | 1 (1)
Blood creatinine increased (Investigations) | 8 (10) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 26 (31)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 (30) | 14 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 8 (11)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 18 (19) | 13 (13)
Leukopenia (Blood and lymphatic system disorders) | 14 (20) | 12 (15)
Increased tendency to bruise (Blood and lymphatic system disorders) | 10 (11) | 7 (7)
Lymphopenia (Blood and lymphatic system disorders) | 18 (27) | 6 (7)
Headache (Nervous system disorders) | 23 (30) | 34 (43)
Dizziness (Nervous system disorders) | 10 (10) | 11 (14)
Tremor (Nervous system disorders) | 10 (11) | 2 (2)
Paraesthesia (Nervous system disorders) | 7 (8) | 9 (10)
Nausea (Gastrointestinal disorders) | 34 (46) | 39 (54)
Diarrhoea (Gastrointestinal disorders) | 24 (31) | 25 (33)
Vomiting (Gastrointestinal disorders) | 21 (27) | 25 (29)
Abdominal pain upper (Gastrointestinal disorders) | 10 (13) | 11 (12)
Constipation (Gastrointestinal disorders) | 11 (11) | 11 (11)
Dyspepsia (Gastrointestinal disorders) | 10 (12) | 5 (6)
Rash (Gastrointestinal disorders) | 13 (17) | 19 (26)
Pruritus (Gastrointestinal disorders) | 10 (11) | 10 (15)
Alopecia (Gastrointestinal disorders) | 12 (12) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 36 (48) | 31 (42)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 37 (47) | 18 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 22 (22) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (25) | 16 (17)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 (13) | 13 (13)
Cushingoid (Endocrine disorders) | 9 (9) | 3 (3)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 20 (21) | 12 (13)
Nasopharyngitis (Infections and infestations) | 30 (46) | 25 (38)
Upper respiratory tract infection (Infections and infestations) | 24 (33) | 24 (28)
Urinary tract infection (Infections and infestations) | 23 (33) | 12 (19)
Pneumonia (Infections and infestations) | 11 (11) | 11 (12)
Sinusitis (Infections and infestations) | 12 (12) | 10 (10)
Bronchitis (Infections and infestations) | 10 (11) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI shall provide Sponsor with an advance copy of any proposed publication or oral presentation at least 60 days prior to the planned date of submission or presentation and Sponsor shall have 60 days to review the proposed publication. Sponsor may request in writing, and the PI shall agree to, (a) the deletion of any Confidential Information, (b) any reasonable changes requested by Sponsor, or (c) a delay of such proposed submission for an additional period, not to exceed 90 days.

DOCUMENTS (2):
  • Study Protocol (2019-01-18): https://cdn.clinicaltrials.gov/large-docs/27/NCT02994927/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT02994927/SAP_001.pdf